CLINICAL TRIAL: NCT07329985
Title: THE EFFECT OF FEAR OF HYPOGLYCEMIA ON DIET AND MEDICATION ADHERENCE IN PATIENTS WITH DIABETES
Brief Title: FEAR of HYPOGLYCEMIA in PATIENTS WITH DIABETES
Status: Not yet recruiting | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Burcu Bayrak3
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Diet, Healthy; Medication Adherence; Hypoglycemia
Keywords: Diabetes; Medication Adherence; Nursing; Diet
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence; Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fear of hypoglycemia has a significant impact on both medication and dietary adherence in individuals with diabetes. Through avoidance behaviors, it can disrupt metabolic control, prevent the achievement of glycemic targets, and increase the risk of long-term complications. Therefore, monitoring only biochemical parameters is insufficient in diabetes management. It is crucial for healthcare professionals to systematically assess the fear of hypoglycemia.

DETAILED DESCRIPTION:
Fear of hypoglycemia can directly affect individuals' adherence to treatment, dietary habits, and self-management behaviors. Low levels of fear can lead to ignoring the risk of hypoglycemia, downplaying symptoms, and creating a predisposition to subsequent hypoglycemic attacks, increasing the risk of life-threatening complications. On the other hand, excessively high levels of fear can create constant anxiety, emotional stress, discomfort, and feelings of insecurity, reducing quality of life and triggering depressive symptoms. Furthermore, individuals with high levels of fear tend to maintain higher glucose levels to avoid hypoglycemia. This leads to impaired metabolic control and an increased risk of long-term complications. Additionally, fear of hypoglycemia can significantly affect how individuals regulate their insulin doses, physical activity, and food intake.The literature indicates that fear of hypoglycemia triggers avoidance behaviors in individuals with diabetes, which often leads to poor treatment adherence. These avoidance behaviors include strategies such as consciously reducing insulin doses, skipping oral antidiabetic medications, or not adhering to the treatment plan. This makes it difficult to reach target glycemic levels, increasing the risk of complications in the long term. Fear of hypoglycemia can negatively affect not only medication adherence but also dietary and nutritional behaviors. It is common for individuals who want to avoid hypoglycemia to consume more carbohydrates than planned meals, add excessive snacks to protect against nocturnal hypoglycemia, or develop irregular eating habits. These behaviors can lead to impaired glycemic control, weight gain, and hyperglycemia, hindering the achievement of metabolic goals. This study aims to address an important gap in diabetes management by examining the impact of fear of hypoglycemia on dietary and medication adherence in patients with diabetes. Fear of hypoglycemia may lead patients to consciously or unconsciously reduce medication doses, skip meals, or deviate from recommended dietary plans. Such behaviors can result in poor glycemic control and increase the risk of diabetes-related complications in the long term. The findings of this study are expected to help healthcare professionals identify fear of hypoglycemia at an early stage and develop individualized education, counseling, and care plans. Consequently, improving treatment adherence and enhancing the quality of life of patients with diabetes may be achieved.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with diabetes Aged 18-65 Having experienced at least one hypoglycemic attack previously, Using antidiabetic medication (oral pills and/or insulin), Volunteered to participate in the study

Exclusion Criteria:

unable to communicate in the same language having cognitive impairment wanting to leave the study at any stage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients who applied to a Training and Research Hospital in Türkiye constituted the study population.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemia Fear Levels in Patients | 15.01.2026-15.06.2025
  The first measure of the study will be the patients' fear of hypoglycemia. The Hypoglycemia Fear Scale will be used for this purpose. The scale score ranges from 0 to 128. While there is no cutoff point for the scale, a higher average score indicates a higher level of fear of hypoglycemia.
Patient Medication Adherence | 15.01.2026-15.06.2025
  The second measure of the study will be patient medication adherence. The Medication Adherence Report Scale will be used for this purpose. Scores on the scale range from 5 to 25. Higher scores indicate adherence, while lower scores indicate non-adherence.
Dietary Adherence of Patients | 15.01.2026-15.06.2025
  Another criterion of the study will be measuring the dietary adherence of the patients. The Mediterranean Diet Adherence Scale will be used for this purpose. A total score of 7 or higher indicates acceptable adherence to the Mediterranean diet, while a score of 9 or higher indicates strict adherence.